CLINICAL TRIAL: NCT02959099
Title: Incident COronary EveNts Identified by Computed Tomography
Acronym: ICONIC
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1310014469
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Atherosclerosis
Keywords: Acute coronary syndrome (ACS); Atherosclerotic plaque morphology; Coronary Computed Tomographic Angiography (CCTA); Gender disparities
MeSH Terms: conditions — Atherosclerosis; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with acute coronary syndrome (ACS).
- Controls: Patients without acute coronary syndrome (ACS).

SUMMARY:
The Incident COronary EveNts Identified by Coronary Tomography (ICONIC) trial is a nested, case-control study derived from the dynamic CONFIRM registry, and is based on propensity scoring methods to match subjects with (cases) or without (controls) acute coronary syndrome (ACS). Our primary objective is to determine CCTA-based atherosclerotic plaque characteristics that would help elucidate precursors of incident ACS, with the secondary objective being an analysis of gender-specific disparities.

DETAILED DESCRIPTION:
Acute myocardial infarctions resulting from unstable plaque in patients with coronary artery disease (CAD) account for a significant portion of cardiovascular morbidity and mortality. Although prediction models that incorporate traditional risk factors have been developed in order to risk stratify patients at highest risk for development of subsequent cardiovascular events, such models lack precision and are often found to over or under-estimate risk. Moreover, current clinical practice has focused on stenosis severity as a predictor of future plaque erosion and/or rupture, in spite of the fact that evidence from intravascular ultrasound (IVUS) studies, such as the PROSPECT trial, demonstrate that ACS events are more likely to occur in less than severely stenotic lesions. Furthermore, there is incomplete understanding of the influence of gender on atherosclerotic plaque composition and downstream coronary events, given the chronologic and prognostic differences between men and women in atherosclerotic cardiovascular disease.

Several studies have attempted elucidating characteristics of vulnerable plaque using invasive imaging modalities such as IVUS. However, such studies have several limitations, most significantly is the fact that plaque characterization was performed after an acute coronary event, which limits the ability to isolate baseline plaque characteristics from changes following the acute event. Noninvasive evaluation of atherosclerotic coronary disease using coronary computed tomographic angiography (CCTA) has been established as an accurate and readily available imaging modality in clinical practice. In addition to the evaluation of diameter stenosis, CCTA is capable of evaluation plaque composition as well as arterial remodeling, in a similar fashion to IVUS. The agreement between plaque characterization using IVUS and CCTA has been demonstrated in several large-scale trials. Nevertheless, there are several key aspects that have yet to be addressed, including the utility of plaque characterization by CCTA for determination of future cardiovascular events, and gender-based differences in atherosclerotic plaque composition in patients with stable and unstable coronary artery disease.

The ICONIC trial was designed as a nested case-control study based on the previously published CONFIRM registry, evaluating demographic, clinical as well as baseline CCTA-determined plaque composition in 238 patients with subsequent ACS events and 238 matched patients without ACS events. As previously described, ICONIC utilizes CCTA to comprehensively assess plaque morphology and characteristics, in addition to arterial wall changes in order to determine characteristics implicated in future adverse events, beyond what has been traditionally described using invasive imaging modalities. The primary goal is to investigate differences in atherosclerotic plaque composition in patients with ACS, compared to patients with stable coronary disease. The secondary goal is to determine gender-specific differences in plaque composition in both stable and unstable coronary artery disease.

ELIGIBILITY:
Cases:

Inclusion criteria:

* Age ≥18 years.
* Adjudicated STEMI / NSTEMI / UA / Unclassified MI (except for type 4a, 4b, or 5 MI)
* Baseline CCTA.

Exclusion criteria:

* Myocardial infarction not meeting the definition of ACS with missing cardiac biomarkers.
* Prior history of CAD (revascularization or MI).
* Prior revascularization (PCI or CABG).
* ACS in a previously revascularized segment.
* Type 4a, 4b, or 5 MI.

Controls

Inclusion criteria:

* Age ≥18 years.
* Propensity score matched.

Exclusion criteria:

* Prior history of CAD (revascularization or MI).
* Death as an outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were recruited from 13 international sites in Asia, Europe and North America, with central adjudication of clinical outcomes and core-laboratory measurement of CCTA-based plaque characteristics.
  Subjects recruited in ICONIC represent individuals suspected of having CAD, meeting the inclusion criteria, and undergoing coronary luminal evaluation using ≥ 64-detector row CCTA. Subjects with established CAD were excluded from the trial. The two arms of the study were patients with baseline CCTA and subsequent occurrence of an ACS event (cases) and patients with baseline CCTA and no subsequent ACS event (controls).
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2012-07-20 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
ACS | within 5 years
  ACS: ST elevation MI (STEMI), non-ST elevation MI (NSTEMI), or unstable angina (UA)

SECONDARY OUTCOMES:
STEMI and NSTEMI | within 5 years
  ST elevation MI (STEMI) or Non-ST elevation MI (NSTEMI)

CONTACTS AND LOCATIONS:
Overall Officials: Leslee J Shaw, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (13):
- United States (3):
  - Baptist Hospital of Miami, Miami, Florida
  - Walter Reed Army Medical Center, Bethesda, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
- Innsbruck Medical University, Innsbruck, Austria
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Providence Health Care St. Paul's Hospital, Vancouver
- University of Munich, Munich, Germany
- Italy (2):
  - Department of Clinical Sciences and Community Health, University of Milan & Centro Cardiologico Monzino, IRCCS, Milan
  - University Hospital of Parma, Parma
- Leiden University Medical Center, Leiden, Netherlands
- Hospital da Luz, Lisbon, Portugal
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Cardiovascular Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Min JK, Dunning A, Lin FY, Achenbach S, Al-Mallah MH, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Cheng V, Chinnaiyan KM, Chow B, Delago A, Hadamitzky M, Hausleiter J, Karlsberg RP, Kaufmann P, Maffei E, Nasir K, Pencina MJ, Raff GL, Shaw LJ, Villines TC. Rationale and design of the CONFIRM (COronary CT Angiography EvaluatioN For Clinical Outcomes: An InteRnational Multicenter) Registry. J Cardiovasc Comput Tomogr. 2011 Mar-Apr;5(2):84-92. doi: 10.1016/j.jcct.2011.01.007. Epub 2011 Feb 1. PMID 21477786
- [Background] Motoyama S, Kondo T, Sarai M, Sugiura A, Harigaya H, Sato T, Inoue K, Okumura M, Ishii J, Anno H, Virmani R, Ozaki Y, Hishida H, Narula J. Multislice computed tomographic characteristics of coronary lesions in acute coronary syndromes. J Am Coll Cardiol. 2007 Jul 24;50(4):319-26. doi: 10.1016/j.jacc.2007.03.044. Epub 2007 Jul 6. PMID 17659199
- [Background] Motoyama S, Sarai M, Harigaya H, Anno H, Inoue K, Hara T, Naruse H, Ishii J, Hishida H, Wong ND, Virmani R, Kondo T, Ozaki Y, Narula J. Computed tomographic angiography characteristics of atherosclerotic plaques subsequently resulting in acute coronary syndrome. J Am Coll Cardiol. 2009 Jun 30;54(1):49-57. doi: 10.1016/j.jacc.2009.02.068. PMID 19555840
- [Background] Pflederer T, Marwan M, Schepis T, Ropers D, Seltmann M, Muschiol G, Daniel WG, Achenbach S. Characterization of culprit lesions in acute coronary syndromes using coronary dual-source CT angiography. Atherosclerosis. 2010 Aug;211(2):437-44. doi: 10.1016/j.atherosclerosis.2010.02.001. Epub 2010 Feb 10. PMID 20189568
- [Background] Cheng VY, Nakazato R, Dey D, Gurudevan S, Tabak J, Budoff MJ, Karlsberg RP, Min J, Berman DS. Reproducibility of coronary artery plaque volume and composition quantification by 64-detector row coronary computed tomographic angiography: an intraobserver, interobserver, and interscan variability study. J Cardiovasc Comput Tomogr. 2009 Sep-Oct;3(5):312-20. doi: 10.1016/j.jcct.2009.07.001. Epub 2009 Jul 30. PMID 19709947
- [Background] Pundziute G, Schuijf JD, van Velzen JE, Jukema JW, van Werkhoven JM, Nucifora G, van der Kley F, Kroft LJ, de Roos A, Boersma E, Reiber JH, Schalij MJ, van der Wall EE, Bax JJ. Assessment with multi-slice computed tomography and gray-scale and virtual histology intravascular ultrasound of gender-specific differences in extent and composition of coronary atherosclerotic plaques in relation to age. Am J Cardiol. 2010 Feb 15;105(4):480-6. doi: 10.1016/j.amjcard.2009.09.054. Epub 2010 Jan 5. PMID 20152242